CLINICAL TRIAL: NCT02704949
Title: Impact of Low Dose Fluoroscopy in Ureteroscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 13788
Record Dates: First submitted 2016-02-17; First posted 2016-03-10 (Estimated); Last update posted 2021-09-29 (Actual); Status verified 2016-02

CONDITIONS: Ureteral Stone
Keywords: Urolithiasis; Fluoroscopy; Radiation; Ureteroscopy
MeSH Terms: conditions — Ureterolithiasis; Urolithiasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low-dose (Experimental): The intervention is to use 1/4 fluoroscopy dose while the ureteroscopy is being performed
  Interventions: Radiation: 1/4 fluoroscopy dose
- Full-dose (Active Comparator): The intervention is to use full fluoroscopy dose while the ureteroscopy is being performed
  Interventions: Radiation: Full-dose

INTERVENTIONS:
Radiation: 1/4 fluoroscopy dose — Use of 1/4 fluoroscopy dose while ureteroscopy is being performed
  Arms: Low-dose
Radiation: Full-dose — Use of full fluoroscopy dose while ureteroscopy is being performed
  Arms: Full-dose

SUMMARY:
One of the most effective strategies to decrease radiation exposure during ureteroscopy is to use low dose. However, the quality of the image obtained is inferior to full dose image. The main concern is to maintain the stone free and complication rate despite the inferior quality of image obtained. Our aim was to evaluate if reducing the dose of fluoroscopy to ¼ instead of full dose would impact in a reduction of total radiation exposure despite a possible increase in fluoroscopy time. Also, if this strategy would impact in operation time, stone free rate and complication rate of unilateral semi-rigid ureteroscopy for ureteral stone treatment due too less than optimal fluoroscopy image. All patients over 18 years old diagnosed with ureteral stone from 5 mm to 20 mm in diameter by CT scan were counseled regarding their treatment options. Patients who failed spontaneous passage or medical treatment or chose endourologic treatment were included in this study. Patients with abnormal urinary anatomy such as horseshoe kidney, pelvic kidney or duplex system were excluded from the study.

DETAILED DESCRIPTION:
Several studies support an association between increasing cancer risk with increasing exposure to radiation. Typical radiation exposure for a patient submitted to ureteroscopy ranges from 2.5 to 100 mSv. The International Commission on Radiological Protection recommends an annual occupational radiation exposure limit of no more than 50 mSv per year. One of the most effective strategies to decrease radiation exposure during ureteroscopy is to use low dose. However, the quality of the image obtained is inferior to full dose image. The main concern is to maintain the stone free and complication rate despite the inferior quality of image obtained. Our aim was to evaluate if reducing the dose of fluoroscopy to ¼ instead of full dose would impact in a reduction of total radiation exposure despite a possible increase in fluoroscopy time. Also, if this strategy would impact in operation time, stone free rate and complication rate of unilateral semi-rigid ureteroscopy for ureteral stone treatment due too less than optimal fluoroscopy image. All patients over 18 years old diagnosed with ureteral stone from 5 mm to 20 mm in diameter by CT scan were counseled regarding their treatment options. Patients who failed spontaneous passage or medical treatment or chose endourologic treatment were included in this study. Patients with abnormal urinary anatomy such as horseshoe kidney, pelvic kidney or duplex system were excluded from the study.

ELIGIBILITY:
Inclusion Criteria:

* ureteral stone from 5 mm to 20 mm in diameter by CT scan

Exclusion Criteria:

* abnormal urinary anatomy such as horseshoe kidney, pelvic kidney or duplex system

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2015-08; Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
radiation exposure | 2 years
  Each group of patients (1/4 dose and full dose) will have assigned one dosimeter to assess the radiation exposure every procedure. The sum of radiation of each group will be compared at the completion of the study (2 years) , because individual radiation exposure is too low to be measured. Radiation exposure will be measured (data stored inside the dosimeter) by dosimeter in mSv units at each procedure and the total sum of radiation will be done at the end of the study (2 years).

SECONDARY OUTCOMES:
stone free rate | 3 months
  None residual fragment in the ureter identified by computed tomography 3 months after the procedure
complications | 3 months
  Clavien-Dindo surgical complication score

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Danilovic, MD, Principal Investigator — University of Sao Paulo General Hospital
Locations (1):
- University of Sao Paulo General Hospital, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No